CLINICAL TRIAL: NCT00972075
Title: A Double-Blind, Placebo-Controlled Study of Circadin™ for Non-24 Hour Sleep-Wake Disorder in Totally Blind Subjects
Brief Title: Efficacy and Safety of Circadin for Non-24 Hour Sleep-Wake Disorder in Totally Blind Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Neurim Pharmaceuticals Ltd. (Industry)
Responsible Party: Tali Nir, VP clinical and regulatory affairs, Neurim Pharmaceuticals Ltd.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CIRCADIN 1
Record Dates: First submitted 2009-09-03; First posted 2009-09-04 (Estimated); Last update posted 2009-09-09 (Estimated); Status verified 2009-09

CONDITIONS: Non-24 Hour Sleep-Wake Disorder; Blindness
Keywords: totally blind subjects
MeSH Terms: conditions — Sleep Disorders, Circadian Rhythm; Blindness | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Circadin (Experimental): Circadin is 2 mg of prolonged release melatonin
  Interventions: Drug: melatonin (Circadin)
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: melatonin (Circadin) — 2 mg prolonged release melatonin tablets once daily 2 hours before going to bed
  Other Names: Circadin; ATC code N05CH01
  Arms: Circadin
Drug: placebo — one tablet per day 2 hours before going to bed
  Arms: Placebo

SUMMARY:
The aim of this placebo-controlled randomized study was to evaluate the efficacy of Circadin™ 2 mg in improving total night sleep duration and stabilizing the circadian clock phase in totally blind subjects with non-24 hour sleep-wake disorder.

DETAILED DESCRIPTION:
This was a multi-center, double-blind, placebo-controlled study of a once-daily (QD) dose of Circadin™ 2 mg in subjects with non-24 hour sleep-wake disorder. Subjects were initially treated with placebo for 2 weeks and then were randomly assigned in a 1:1 ratio to receive Circadin™ 2 mg or placebo for 6 weeks, followed by a 2-week washout period. The primary objective was to assess the effect of Circadin 2 mg given once daily for 6 weeks on total night sleep duration. Secondary objectives were other sleep variables recorded by the diary like sleep latency, daytime naps and sleep offset time. Other endpoints were CGIC score for Severity of Illness and Global Improvement and WHO (Five) Well-Being Index score.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged 20-80, having no conscious perception of light.
* Meeting the criteria for diagnosing Non-24h cycle in the clinical setting: 1) difficulty initiating sleep or difficulty in awakening, 2) progressive delay of sleep phase with inability to maintain entrainment to 24-hour-day, and 3) presence of the sleep pattern for at least six weeks.
* Average total night sleep duration of less than 6 hours per night for at least six weeks.
* Ability to ingest oral medication and participate in all scheduled evaluations.
* Signing of the Informed Consent approved by the Ethics Committee. The Informed Consent will be written in both Braille and black-and-white forms for blind subject and sighted witness.
* Education or a work history sufficient to exclude mental retardation.
* Stable medications for non-excluded concurrent medical conditions for four weeks prior to the screening visit.

Exclusion Criteria:

* Presence of medical disorders other than those related to blindness and medical treatment that may influence melatonin production, sleep or alertness. To be ascertained by medical history, complete physical examination including ECG and general biochemical work-up including complete blood count, serum chemistries, and urine analysis.
* Presence of a psychiatric or mental disorder to be assessed by a structured psychiatric interview performed by a trained individual.
* History of seizure disorders.
* Irregular lifestyle or life pattern (e.g. shift workers and patients unable to keep the study routine).
* Presence of a sleep problem revealed that may explain the subjects' complaints, such as sleep disordered breathing, restless leg syndrome or periodic limb movement syndrome.
* Use of benzodiazepines or other hypnotics during the study and preceding two weeks or 5 half lives whichever is longer.
* Known or suspected hypersensitivity to exogenous melatonin or melatonin receptor agonists
* Use of melatonin during preceding two weeks
* Use of psychiatric medications during the study and preceding three months.
* History of autoimmune diseases
* Pharmacological immuno-suppression.
* Pregnancy or lactation, child-bearing potential with a lack of adequate contraception.
* History of severe pathology likely to recur during or immediately after the study.
* Participation in a clinical trial with any investigational agent within two months prior to study enrollment.
* Patients incapable of performing the daily call to the study IVRS system and reporting on the questionnaires.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2006-02; Primary Completion 2007-08 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Total sleep time | six weeks

SECONDARY OUTCOMES:
Daily diary records of sleep latency, sleep maintenance , total duration of naps; | six weeks

CONTACTS AND LOCATIONS:
Overall Officials: Alan Lankford, PhD, Principal Investigator — Sleep Disorders Center of Atlanta; Gary Zammit, PhD, Principal Investigator — Clinlabs, Inc.
Locations (2):
- United States (2):
  - Sleep Disorders Center of Atlanta, Atlanta, Georgia
  - Clinlabs, Inc., New York, New York

REFERENCES:
- [Derived] Roth T, Nir T, Zisapel N. Prolonged release melatonin for improving sleep in totally blind subjects: a pilot placebo-controlled multicenter trial. Nat Sci Sleep. 2015 Jan 29;7:13-23. doi: 10.2147/NSS.S71838. eCollection 2015. PMID 25678831